CLINICAL TRIAL: NCT00826267
Title: Randomised Phase II Study of Neoadjuvant BIBW 2992 Versus Herceptin Versus Lapatinib in Her2 Positive Breast Cancer Patients
Brief Title: 6 Weeks Treatment of Locally Advanced Breast Cancer With BIBW 2992 (Afatinib) or Lapatinib or Trastuzumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200.44
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-08

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Afatinib; Trastuzumab

ARMS (3):
- BIBW 2992 (Experimental): BIBW 2992 high dose once daily (allowed dose reduction to medium or low once daily in case of AE)
  Interventions: Drug: BIBW 2992
- Lapatinib (Active Comparator): Lapatinib tablets 1500 mg daily.
  Interventions: Drug: lapatinib
- Trastuzumab (Active Comparator): Trastuzumab 4mg/kg i.v. week 1, followed by 2mg/kg i.v. weekly.
  Interventions: Drug: trastuzumab

INTERVENTIONS:
Drug: lapatinib — lapatinib tablets 1500 mg daily
  Arms: Lapatinib
Drug: BIBW 2992 — BIBW 2992 high dose once daily (allowed dose reduction to medium or low once daily in case of AE)
  Arms: BIBW 2992
Drug: trastuzumab — trastuzumab 4mg/kg i.v. week 1, followed by 2mg/kg i.v. weekly
  Arms: Trastuzumab

SUMMARY:
An open-label, randomized three-arm Phase II trial to explore the efficacy of BIBW 2992 as a single agent versus lapatinib versus trastuzumab in patients with HER2-positive treatment-naïve Stage IIIa locally advanced breast cancer. Additional information will be obtained on the safety profile and pharmacokinetics of BIBW 2992.

ELIGIBILITY:
Inclusion criteria:

1. Female, age 18 years or older.
2. Histologically proven breast cancer who have not received any prior therapy.
3. Locally advanced disease Stage IIIa with no evidence of distant metastatic disease other than anatomical site lymph nodes.
4. HER2-positive.

Exclusion criteria:

1. Absolute neutrophil count (ANC) less than 1500/mm3.
2. Platelet count less than 100 000/ mm3.
3. Hemoglobin level less than 9.0 g/dl.
4. Bilirubin greater than 1.5 mg/dI.
5. Aspartate amino transferase (AST) or alanine amino transferase (ALT) greater than twice the upper limit of normal.
6. Serum creatinine greater than 1.5 times of the upper normal limit.
7. Significant or recent acute gastrointestinal disorders with diarrhea
8. Pregnancy or breast-feeding.
9. Organ system dysfunction including cardiac (LVEF < 50%).
10. Prior chemotherapy, radiotherapy or hormone therapy. Previous treatment with trastuzumab, EGFR, or EGFR/HER2-inhibitors.
11. Other malignancies diagnosed within the past five years.
12. Serious active infection. HIV, active hepatitis B or C.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-01; Primary Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (17):
- 1200.44.01001 Boehringer Ingelheim Investigational Site, Houston, Texas, United States
- Brazil (10):
  - 1200.44.12008 Boehringer Ingelheim Investigational Site, Brasília
  - 1200.44.12011 Boehringer Ingelheim Investigational Site, Cachoeiro de Itapemirim
  - 1200.44.12012 Boehringer Ingelheim Investigational Site, Campo Grande
  - 1200.44.12009 Boehringer Ingelheim Investigational Site, Caxias do Sul
  - 1200.44.12010 Boehringer Ingelheim Investigational Site, Goiânia
  - 1200.44.12005 Boehringer Ingelheim Investigational Site, Ijuí
  - 1200.44.12007 Boehringer Ingelheim Investigational Site, Natal
  - 1200.44.12004 Boehringer Ingelheim Investigational Site, Novo Hamburgo
  - 1200.44.12001 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1200.44.12013 Boehringer Ingelheim Investigational Site, Porto Alegre
- Colombia (2):
  - 1200.44.14002 Boehringer Ingelheim Investigational Site, Bogotá
  - 1200.44.14001 Boehringer Ingelheim Investigational Site, Cali
- Peru (4):
  - 1200.44.19005 Boehringer Ingelheim Investigational Site, Cercado
  - 1200.44.19001 Boehringer Ingelheim Investigational Site, Lima
  - 1200.44.19004 Boehringer Ingelheim Investigational Site, Lima
  - 1200.44.19003 Boehringer Ingelheim Investigational Site, San Isidro

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Because of slow enrollment and a high screen-failure rate, recruitment became a challenge and the sponsor chose to terminate the trial prior to reaching the target enrollment of 120 patients.
Groups:
- Afatinib 50 mg: Patients received continuous daily dosing with Afatinib 50 mg orally from Day 1 to Day 21 of each treatment course. 2 treatment courses were to be given in the trial.
- Lapatinib 1500 mg: Patients received continuous daily dosing with Lapatinib 1500 mg orally from Day 1 to Day 21 of each treatment course. 2 treatment courses were to be given in the trial.
- Trastuzumab: Patients received weekly trastuzumab infusions of 2 mg/kg following a loading dose of 4 mg/kg per SPC. 6 infusions were to be given over 2 treatment courses.
Period: Overall Study
Arm/Group | Afatinib 50 mg | Lapatinib 1500 mg | Trastuzumab
Started | 10 | 8 | 11
Completed | 9 | 8 | 11
Not Completed | 1 | 0 | 0
Not completed — Other Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib 50 mg | Lapatinib 1500 mg | Trastuzumab | Total
Number analyzed (Participants) | 10 | 8 | 11 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (8.7) | 58.5 (13.4) | 44.1 (12.2) | 50.3 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 11 | 29
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (OR)
Description: Objective response (complete or partial) was assessed according to RECIST 1.0 criteria.
Time Frame: Tumour assessments were performed at screening, day 22 and day 43.
Population: Treated set (TS). TS consisted of all patients who received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib 50 mg | Lapatinib 1500 mg | Trastuzumab
Number analyzed (Participants) | 10 | 8 | 11
Percentage of participants | 80.0 [44.4 to 97.5] | 75.0 [34.9 to 96.8] | 36.4 [10.9 to 69.2]

2. Secondary Outcome: Number of Participants Who Achieved Clinical Benefit (CB)
Description: CB was defined as CR, PR or stable disease (SD) and was assessed according to RECIST criteria regardless of treatment status.
Time Frame: Tumour assessments were performed at screening, day 22 and day 43.
Population: TS
Measure: Number; unit: Participants
Arm/Group | Afatinib 50 mg | Lapatinib 1500 mg | Trastuzumab
Number analyzed (Participants) | 10 | 8 | 11
Participants | 10 | 8 | 11

3. Secondary Outcome: Change From Baseline in the Diameter of the Primary Target Lesion.
Description: Change was based on the primary lesion only rather that the sum of the target lesions as most patients had only one lesion.
Time Frame: 3 weeks or 6 weeks
Population: TS
Measure: Least Squares Mean (Standard Error); unit: millimeters
Arm/Group | Afatinib 50 mg | Lapatinib 1500 mg | Trastuzumab
Number analyzed (Participants) | 10 | 8 | 11
millimeters | -27.5 (5.90) | -31.0 (6.63) | -20.9 (5.63)

4. Secondary Outcome: Plasma Concentration of Afatinib
Description: Individual drug plasma concentrations of afatinib after multiple oral administrations at day 7
Time Frame: Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Afatinib 50mg: Patients received Afatinib 50 mg at day 7.
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 10
ng/mL | 32.1 (43.0)

5. Secondary Outcome: Changes in Biomarker in Tumour Biopsies
Description: Changes in the biomarkers (Phospho-MAP-Kinase (MAPK), Total MAPK expression, EGFR, HER2, Phospho-EGFR and -HER2, Proliferation marker (Ki67 and p27), Apoptotic index (cleaved caspase 3), Phosphate and tensin homolog (PTEN), HER2 homodimerisation by HERmark assay and Phospho AKT) from biopsy tissue.
Time Frame: Screening, day 22, day 43
Population: TS. The small number of available biomarker samples in this study did not allow for a meaningful statistical analysis.
Arm/Group | Afatinib 50 mg | Lapatinib 1500 mg | Trastuzumab
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 28 days following the end-of-treatment visit.
Arm/Group | Afatinib 50 mg | Lapatinib 1500 mg | Trastuzumab
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 10/10 | 8/8 | 8/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 50 mg (N=10) | Lapatinib 1500 mg (N=8) | Trastuzumab (N=11)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphatic disorder (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Cyanosis (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 10 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 3
Oral discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2
Asthenia (General disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 2
Fatigue (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Mucosal inflammation (General disorders) | 4 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Paronychia (Infections and infestations) | 5 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Viral sinusitis (Infections and infestations) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 4
Tremor (Nervous system disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 6 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Because of slow enrollment and a high screen-failure rate, recruitment became a challenge and the sponsor chose to terminate the trial prior to reaching the target enrollment of 120 pat. Small number of subjects lead to some shortcomings in analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.